CLINICAL TRIAL: NCT02353260
Title: A Randomized Controlled Clinical Trial to Evaluate the Efficacy and Safety of Ultrasound Hyperthermia in Combination With Chemotherapy on Oral and Maxillofacial-Head and Neck Cancer
Brief Title: Efficacy and Safety of Ultrasound Hyperthermia Combined With Chemotherapy on Oral and Maxillofacial-Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Guo (Other)
Collaborators: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Wei Guo, Director in Dept.of Oral and Maxillofacial-Head and Neck Oncology, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-A
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; CF regimen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound Hyperthermia+Chemotherapy (Experimental): Chemotherapy:
  1. Squamous cell carcinoma of head and neck: Docetaxel(75mg/m²,d1/21d,2 cycles);Cisplatin(75mg/m²,d1/21d,2 cycles);Fluorouracil(750mg/m²/d,d1-5/21d, 2 cycles)
  2. The treatments will be administrated in accord with the guideline for other types of cancer.
  Ultrasound Hyperthermia: Ultrasound hyperthermia d1,3,5,7,9/21d for 2 cycles
  Interventions: Device: Ultrasound Hyperthermia; Drug: Docetaxel,Cisplatin,Fluorouracil
- Chemotherapy (Active Comparator): Chemotherapy:
  1. Squamous cell carcinoma of head and neck: Docetaxel(75mg/m²,d1/21d,2 cycles);Cisplatin(75mg/m²,d1/21d,2 cycles);Fluorouracil(750mg/m²/d,d1-5/21d, 2cycles)
  2. The treatments will be administrated in accord with the guideline for other types of cancer.
  Interventions: Drug: Docetaxel,Cisplatin,Fluorouracil

INTERVENTIONS:
Device: Ultrasound Hyperthermia — treated with Therapeutic Ultrasound device on the 1st,3rd,5th,7th,9th day of each 21 day cycle
  Arms: Ultrasound Hyperthermia+Chemotherapy
Drug: Docetaxel,Cisplatin,Fluorouracil — Squamous cell carcinoma of head and neck: Docetaxel(75mg/m²,d1/21d,2 cycles);Cisplatin(75mg/m²,d1/21d,2 cycles);Fluorouracil(750mg/m²/d,d1-5/21d, 2 cycles)

SUMMARY:
The purpose of this study is to determine whether Ultrasound Hyperthermia is effective and safe in the treatment of Oral and Maxillofacial-Head and Neck Cancer.

DETAILED DESCRIPTION:
As a non-invasive treatment, Ultrasound Hyperthermia has received increasing interest for the treatment of cancer.Many studies have shown that Therapeutic Ultrasound is safe and effective. Eligible patients were randomly assigned by using permutated blocks designed for each site to receive either Ultrasound Hyperthermia combined with chemotherapy (Arm A) or chemotherapy alone(Arm B).Chemotherapy will be conducted as follows. For Squamous cell carcinoma of head and neck,it will be administrated with Docetaxel(at a dose of 75 mg per square meter of body-surface area and intravenous infused in 1 hr at day 1rt), Cisplatin(at a dose of 75 mg per square meter of body-surface area and intravenous infused in 1 hr at day 1rt) and Fluorouracil(at a dose of 75 mg per square meter of body-surface area and intravenous infused last 5 days) . For other types of cancer,the treatments will be administrated in accord with the guideline.In addition,Ultrasound Hyperthermia will be conducted 5 times(day 1rt,3rd,5th,7th,9th) in Arm A. Patients in arm B will receive chemotherapy only. One cycle comprises a period of 3 weeks (21 days).All patients will receive 2 cycles in both arms. All the patients eligible for the operation will take surgery. After treatment，some patients with advanced unresectable cancer may be down-staged from stage IV, and will regain the opportunity of operation.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntary and signed informed consent form
* Age 18-75，both genders.
* Had histologically or cytologically confirmed advanced squamous cell carcinoma of the head and neck
* At least one lesions can be measured,Conventional measurements ≥2cm, computed tomography(CT) examination ≥1cm .
* Eastern Cooperative Oncology Group(ECOG) Performance Scale 0-2.
* Life expectancy of more than 6 months.
* Use of an effective contraceptive method for women when there is a risk of pregnancy during the study.
* Haemoglobin≥90g/L ,White blood cell(WBC) ≥3×10^9/L
* Hepatic function:ALAT、ASAT< 2.5 x ULN, TBIL< 1.5 x ULN
* Renal function: Creatinine < 1.5 x ULN

Exclusion Criteria:

* Participation in other interventional clinical trials within 1 month
* Previous received other drug or operative treatment within 6 month
* Pregnant or breast-feeding women
* History of serious allergic or allergy
* Patients with the history of Serious lung or head disease
* Local skin ulceration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Disease Control | one year

SECONDARY OUTCOMES:
Progression Free Survival | three years
Over Survival | three years

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, PhD, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China